CLINICAL TRIAL: NCT01676155
Title: The Role of Apoptosis Associated Markers in Pathogenesis of Pulmonary Tuberculosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20110822RC
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-06

CONDITIONS: To Compare the Serum Apoptosis-associated Markers Between Patients With Active TB and Patients With LTBI; To Evaluate the Efficiency of Apoptosis-associated Markers to Differentiate Potential of Active TB From LTBI
Keywords: Tuberculosis, latent tuberculosis infection, apoptosis, predictor
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patient with active tuberculosis
- Patients with diagnosis of latent tuberculosis infection
- Patient without latent tuberculosis or active tuberculosis

SUMMARY:
To compare the serum apoptosis-associated markers between patients with active TB and patients with LTBI To evaluate the efficiency of apoptosis-associated markers to differentiate potential of active TB from LTBI

DETAILED DESCRIPTION:
Background: Tuberculosis (TB) remains the most important infectious disease worldwide. For controlling TB, the important strategy includes not only adequate anti-tuberculous treatment but also well control of latent TB infection (LTBI). Latent TB infection (LTBI) has 10% of reactivation or more in patients with immuno-compromised disorder. Although LTBI can be detected by interferon-gamma release assay (IGRA) or tuberculin skin test, how to predict who will become active TB from LTBI is still unclear but important. In overall prophylactic treatment for LTBI, the lengthy duration and possible serious side effect too scared to general application especially 90% of population who may not get illness. Therefore, to recognize who develop active TB from LTBI is important for targeted prophylactic therapy. The good marker is not discovered at present. When TB bacilli arrive our lung, macrohage is the first line defense and necrosis rather than apoptosis is the dominant form of cell death, which affords a protective milieu for M. tuberculosis. Though the apoptosis is suppressed in TB, the apoptosis-associated markers have rarely been investigated in human LTBI vs. active TB. We set up a cohort study to detect active TB developing from LTBI and first-step conduct a case control study to compare apoptosis markers between LTBI and active TB for evaluating the apoptosis markers in discriminating TB infection status. The significant markers should be verified in further cohort study of LTBI patients.

Hypothesis: The apoptosis-associated markers, including Fas ligand, Decoy-receptor 3, Lipoxin, and prostaglandin E2, are discriminative in patients with active TB from those with LTBI and thus might predict the potential of being active TB from LTBI.

Study Aims:

To compare the serum apoptosis-associated markers between patients with active TB and patients with LTBI To evaluate the efficiency of apoptosis-associated markers to differentiate potential of active TB from LTBI Methods: We prospectively enroll patients with active TB (n=100) and LTBI (n=100), defined by IGRA. Blood sample would be collected before they received definite treatment after yielding informed consent. We will examine serum apoptosis-associated markers including Fas ligand, Decoy-receptor 3, Lipoxin, and prostaglandin E2, and other cytokines and chemokines in serum sample and supernatant from T-cell after TB antigen stimulation. Their clinical characteristics will be recorded. We compare the laboratory and clinical data between the two groups and analyze the efficacy of diagnostic help from these markers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years
* Latent TB group: family contacts who have positive response in IGRA (by QuantiFeron-TB Gold-in-Tube, which is described detail in Part C) and have no signs of active TB.
* Active TB group: patients with pulmonary tuberculosis diagnosed by positive respiratory culture.

Exclusion Criteria:

* Age younger than 20 years.
* Patients who have pregnancy.
* Patients who have acquired immunodeficiency syndrome
* Patients who have bleeding tendency which can not tolerate venous puncture such as hemophilia, thrombocytopenia.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Patients with tuberculosis: microbiology or pathology proven tuberculosis infection
  2. Patients with latent tuberculosis infection are defined by interferon-gamma release assay
  3. Patients without tuberculosis and latent tuberculosis are defi=ed by negative findings in above-mentioned results
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2011-09

PRIMARY OUTCOMES:
getting active tuberculosis | 2 year

SECONDARY OUTCOMES:
mortality | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Chung Shu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan